CLINICAL TRIAL: NCT03216577
Title: Short and Long-term Outcomes of Purpura Fulminans in Adults
Brief Title: Outcomes of Purpura FULminans in Adults - The hOPeFUL Study
Acronym: hOPeFUL
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Principal Investigator, Nicolas de Prost, MD, PhD, Henri Mondor University Hospital
Other Study IDs: hOPeFUL
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Purpura Fulminans
Keywords: health-related quality of life
MeSH Terms: conditions — Purpura Fulminans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to purpura fulminans: Patients who were admitted in the intensive care unit and survived a purpura fulminans episode
  Interventions: Other: Phone interview measuring health-related quality of life variables
- Non-exposed to purpura fulminans: Patients admitted in the intensive care unit for a septic shock unrelated to a purpura fulminans, and matched to exposed patients for age, gender, and severity of illness.
  Interventions: Other: Phone interview measuring health-related quality of life variables

INTERVENTIONS:
Other: Phone interview measuring health-related quality of life variables — A phone interview will be conducted by a dedicated nurse who will be blinded to the exposed/non-exposed status of the patient.

SUMMARY:
Purpura fulminans (PF) is a rare life-threatening infectious disease characterized by the association of a sudden and extensive purpura together with acute circulatory failure. The mortality of PF has been reported to be as high as 50% in previous adult series. Additionally, patients surviving to the early phase of PF are exposed to a high risk of limb amputation. The hOPeFUL study aims at assessing the short and long term outcomes of adult patients admitted in the intensive care unit for a purpura fulminans.

DETAILED DESCRIPTION:
Purpura fulminans (PF) is a rare life-threatening infectious disease characterized by the association of a sudden and extensive purpura together with acute circulatory failure. Neisseria meningitidis and Streptococcus pneumoniae are the most frequently involved microorganisms but other species (e.g., Staphylococcus aureus, Streptococcus pyogenes, Haemophilus influenzae…) have also been reported. Despite prompt antibiotics administration and intensive care management, the mortality of PF has been reported to be as high as 50% in previous adult series. Additionally, patients surviving to the early phase of PF are exposed to a high risk of serious sequelae related to extensive skin necrosis and acral symmetrical gangrene, which typically requires limb amputations, a potential source of severe handicap in these previously young and healthy patients. Although the clinical features and outcomes of PF have been well studied in the pediatric setting, the amount of available data for adult PF are scarce, often outdated and mainly limited to patients with meningococcal infections. The current study aims at assessing the short and long-term outcomes of adult patients admitted in the intensive care unit for a purpura fulminans. A large multicenter retrospective cohort will be built in order to assess hospital outcomes (i.e., mortality and amputations). Long-term outcomes, including health-related quality variables, will be prospectively assessed among survivors and compared to septic controls (i.e., patients having septic shock non-related to purpura fulminans).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the intensive care unit between 2010 and 2016 for an infectious purpura fulminans and discharged alive

Exclusion Criteria:

* Age < 18 years
* Non infectious purpura
* Infective endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in the intensive care unit between 2010 and 2016 for an infectious purpura fulminans (cases/exposed patients) and discharged alive will be matched (gender, age and SAPS II score) to patients admitted during the same time frame for a septic shock non-related to purpura fulminans (controls/non-exposed pâtients).
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | day 60
  factors associated with hospital mortality (and rate of amputation in the hospital) will be identified using a polytomous logistic regression model
Rate of amputation in the hospital; | day 60
  factors associated with rate of amputation in the hospital (and hospital mortality) will be identified using a polytomous logistic regression model
Long-term outcome measure: Physical dimension scale of the SF-36 questionnaire | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans and patients with septic shock non-related to purpura fulminans

SECONDARY OUTCOMES:
Mental component score of the SF-36 score | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans and patients with septic shock non-related to purpura fulminans
Activity of daily living (ADL score) | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans and patients with septic shock non-related to purpura fulminans
Hospital anxiety and depression scale | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans and patients with septic shock non-related to purpura fulminans
Impact of Event Scale | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans and patients with septic shock non-related to purpura fulminans
Physical dimension scale of the SF-36 questionnaire | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans who were and those who were not amputated
Mental component score of the SF-36 score | Within 6 years of hospital discharge
  This variable will be compared between patients with purpura fulminans who were and those who were not amputated

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas de Prost, MD, PhD, Principal Investigator — Henri Mondor University Hospital
Locations (26):
- France (26):
  - Aulnay sous Bois Hospital, Aulnay-sous-Bois
  - Caen University Hospital, Caen
  - Chartres Hospital, Chartres
  - Louis Mourier Hospital, Colombes
  - Henri Mondor Hospital, Créteil
  - Grenoble University Hospital, Grenoble
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Versailles Hospital, Le Chesnay
  - Le Havre Hospital, Le Havre
  - Lilles University Hospital, Lilles
  - Edouard Herriot Hospital, Lyon
  - Melun Hospital, Melun
  - Nice University Hospital, Nice
  - Orléans Hospital, Orléans
  - Saint Louis Hospital, Paris
  - Saint-Antoine Hospital, Paris
  - Pitié-Salpétrière Hospital, Paris
  - Cochin Hospital, Paris
  - Bichat University Hospital, Paris
  - Poissy Hospital, Poissy
  - Poitiers University Hospital, Poitiers
  - Clinique Gallien, Quincy-sous-Sénart
  - Reims University Hospital, Reims
  - Rennes University Hospital, Rennes
  - Roubaix Hospital, Roubaix
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Giraud T, Dhainaut JF, Schremmer B, Regnier B, Desjars P, Loirat P, Journois D, Lanore JJ. Adult overwhelming meningococcal purpura. A study of 35 cases, 1977-1989. Arch Intern Med. 1991 Feb;151(2):310-6. PMID 1992958
- [Result] Lerolle N, Carlotti A, Melican K, Aubey F, Pierrot M, Diehl JL, Caille V, Hekimian G, Gandrille S, Mandet C, Bruneval P, Dumenil G, Borgel D. Assessment of the interplay between blood and skin vascular abnormalities in adult purpura fulminans. Am J Respir Crit Care Med. 2013 Sep 15;188(6):684-92. doi: 10.1164/rccm.201302-0228OC. PMID 23924269
- [Derived] Contou D, Canoui-Poitrine F, Coudroy R, Preau S, Cour M, Barbier F, Terzi N, Schnell G, Galbois A, Zafrani L, Zuber B, Ehrmann S, Gelisse E, Colling D, Schmidt M, Jaber S, Conia A, Sonneville R, Colin G, Guerin L, Roux D, Jochmans S, Kentish-Barnes N, Audureau E, Layese R, Alves A, Ouedraogo R, Brun-Buisson C, Mekontso Dessap A, de Prost N; Hopeful Study Group. Long-term Quality of Life in Adult Patients Surviving Purpura Fulminans: An Exposed-Unexposed Multicenter Cohort Study. Clin Infect Dis. 2019 Jul 2;69(2):332-340. doi: 10.1093/cid/ciy901. PMID 30335142
- [Derived] Contou D, Sonneville R, Canoui-Poitrine F, Colin G, Coudroy R, Pene F, Tadie JM, Cour M, Beduneau G, Marchalot A, Guerin L, Jochmans S, Ehrmann S, Terzi N, Preau S, Barbier F, Schnell G, Roux D, Leroy O, Pichereau C, Gelisse E, Zafrani L, Layese R, Brun-Buisson C, Mekontso Dessap A, de Prost N; Hopeful Study Group. Clinical spectrum and short-term outcome of adult patients with purpura fulminans: a French multicenter retrospective cohort study. Intensive Care Med. 2018 Sep;44(9):1502-1511. doi: 10.1007/s00134-018-5341-3. Epub 2018 Aug 20. PMID 30128591